CLINICAL TRIAL: NCT03187301
Title: A Phase 2, Randomized, Double-Blind, Placebo Controlled, 3-Period Crossover, Positive Control, QT-Evaluation Study of APL-130277 in Subjects With Parkinson's Disease Complicated by Motor Fluctuations ("OFF" Episodes)
Brief Title: A Cardiac Safety Study of an Investigational Drug to See How if Affects the Heart in People With Parkinson's Disease Complicated by Motor Fluctuations "OFF" Episodes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTH-201; 2016-001762-29 (EudraCT Number)
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Parkinson's Disease; Off Episodes of Parkinson Disease
Keywords: Parkinson's Disease; Off episodes
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- APL-130277 (Experimental): APL-130277 at the dose determined in the dose titration phase
  Interventions: Drug: APL-130277
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- moxifloxacin (Active Comparator): moxifloxacin at a single 400mg dose
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: APL-130277 — APL-130277 single dose
  Arms: APL-130277
Drug: Placebo — Placebo single dose
  Arms: Placebo
Drug: Moxifloxacin — moxifloxacin 400mg single dose
  Arms: moxifloxacin

SUMMARY:
A cardiac safety study of an investigational drug to see how it affects the heart in people with Parkinson's Disease Complicated by Motor Fluctuations ("OFF" Episodes)

DETAILED DESCRIPTION:
This multi-center, Phase 2, Randomized, Double-Blind, Placebo Controlled, 3-Period Crossover, Positive Control study designed to evaluate the QT interval prolongation potential of 10 mg to 60 mg doses of APL-130277 compared to placebo and the positive control, 400mg moxifloxacin in subjects with Parkinson's Disease (PD) who experience motor fluctuations ("OFF" episodes) The patient is titrated to the highest tolerated dose from 10mg to 60mg, and then is randomized to one of six crossover sequences. Each sequence includes treatment with the following:

1. Treatment A: APL-130277 at the dose determined in the Dose Titration Phase,
2. Treatment B: Matched placebo,
3. Treatment C: A single 400 mg dose of moxifloxacin

ELIGIBILITY:
Inclusion Criteria:

* 1) Male or female ≥ 18 years of age. 2) Clinical diagnosis of Idiopathic PD, consistent with UK Brain Bank Criteria (excluding the "more than one affected relative" criterion).

  3) Clinically meaningful response to Levodopa (L-Dopa). Subjects with or without well defined "OFF" episodes, as determined by the Investigator will be allowed.

  4) Receiving stable doses of L-Dopa/carbidopa (immediate or sustained release) administered at least 3 times per day OR Rytary™ administered 3 times per day, for at least 4 weeks before the initial Screening Visit (SV1). Subjects receiving L-Dopa/carbidopa 3 times a day must also be on stable treatment with adjunctive PD medication regimens. These regimens bust me maintained at a stable dose for at least 4 weeks prior to the initial Screening Visit (SV1) with the exception that MAO-B inhibitors must be maintained at a stable level for at least 8 weeks prior to the initial Screening Visit (SV1).

  5) No planned medication change(s) or surgical intervention anticipated during the course of study.

  6) the subject must be able to have a drug withdrawal induced "OFF" episode.

  7) Stage III or less on the modified Hoehn and Yahr scale in the "ON" state.

  8) Mini-Mental State Examination (MMSE) score > 21.

  9) If female and of childbearing potential, must agree to use one of the following methods of birth control throughout the study and until at least 30 days after final drug administration:
  * Oral contraceptive
  * Contraceptive patch
  * Barrier (diaphragm, sponge or condom) plus spermicidal preparations
  * Intrauterine contraceptive system
  * Levonorgestrel implant
  * Medroxyprogesterone acetate contraceptive injection
  * Complete abstinence from sexual intercourse;
  * Hormonal vaginal contraceptive ring; or
  * Surgical sterilization or partner sterile (must have documented proof).

    10)Male subjects must be either surgically sterile, agree to be sexually abstinent or use a barrier method of birth control (e.g., condom) from first study drug administration until at least 30 days after final drug administration

    11)Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study-related procedures to complete the study.

    12)Able to understand the consent form, and to provide written informed consent.

    13)Must be approved as a satisfactory candidate by the Enrollment Authorization Committee (EAC) and the Sponsor.

Exclusion Criteria:

1. Atypical or secondary parkinsonism
2. Nausea associated with the use of dopamine agonists that requires treatment with an antiemetic.
3. Previous treatment with any of the following: a neurosurgical procedure for PD; continuous subcutaneous (s.c.) apomorphine infusion; or Duodopa/Duopa.
4. Treatment with any form of s.c. apomorphine within 7 days prior to the initial Screening Visit (SV1). Subjects that stopped s.c. apomorphine for any reason other than systemic safety concerns or lack of efficacy may be considered.
5. Contraindications to moxifloxacin or APOKYN®, or hypersensitivity to apomorphine hydrochloride or any macrolide antibiotic or any of the ingredients of APOKYN® (notably sodium metabisulfite).
6. Female who is pregnant or lactating.
7. Participation in a clinical trial within 30 days prior to the initial Screening Visit (SV1), with the exception of clinical studies related to APL-13077.
8. Receipt of any investigational (i.e., unapproved) medication within 30 days prior to the initial Screening Visit (SV1), with the exception of APL-13077.
9. Any selective 5HT3 antagonists (i.e., ondansetron, granisetron, dolasetron, palonosetron, alosetron), dopamine antagonists (including Tigan [trimethobenzamide] and domperidone, but excluding quetiapine or clozapine) or dopamine depleting agents within 30 days prior to initial Screening Visit (SV1).
10. Drug or alcohol dependency in the past 12 months.
11. Subject has a history of malignancy within 5 years prior to SV1, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. Pituitary tumors of any duration are excluded.
12. Documented abnormalities with ECGs including, arrhythmias, clinically meaningful interval irregularities, structural heart abnormalities ,myocardial infarction, presence or history of a pacemaker, or any abnormality of the ECG that in the opinion of the Investigator, would interfere with the ability to measure the QT interval, or correct the QT interval for heart rate.
13. Male subjects with a screening corrected QT interval using Fridericia's formula (QTcF) of ≥ 450 ms; female subjects with a screening QT interval ≥ 470 ms. Eligibility will be based on the core laboratory ECG interpretation report.
14. HR at screening < 45 bpm or > 100 bpm.
15. QRS duration at screening >120 ms
16. PR interval at screening >200 ms.
17. Subjects with a history of cataplexy, unexplained syncope or seizures.
18. Family history of sudden cardiac death.
19. Heart failure (NYHA Class II or greater) and/or a myocardial infarction.
20. Current use of any concomitant mediations that prolong the QT/QTc interval. Refer to https://crediblemeds.org for listing.
21. History of additional risk factors for TdP (i.e., heart failure, hypokalemia, family history of Long QT Syndrome).
22. Clinically significant medical, surgical, or laboratory abnormality in the opinion of the Investigator.
23. Subject has a positive screening laboratory test result for human immunodeficiency virus (HIV).
24. Subject has a positive screening laboratory test result for hepatitis B surface antigen or hepatitis C antibodies and has liver function test results at screening above the ULN for the reference laboratory.
25. Major psychiatric disorder including, but not limited to, dementia, bipolar disorder, psychosis (including Parkinson's disease psychosis), or any disorder that, in the opinion of the Investigator, requires ongoing treatment that would make study participation unsafe or make treatment compliance difficult.
26. History of clinically significant impulse control disorder(s).
27. Dementia that precludes providing informed consent or would interfere with participation in the study.
28. Current suicidal ideation within one year prior to the second Screening Visit (SV2) as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) or attempted suicide within the last 5 years.
29. Donation of blood plasma in the 30 days prior to first dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Chair — Sunovion Pharmacetuicals Inc.
Locations (15):
- United States (10):
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - MD Clinical, Hallandale, Florida
  - Bioclinica Reserach, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - The NeuroMedical Center, PC, Baton Rouge, Louisiana
  - QUEST Research Institute, Farmington Hills, Michigan
  - Central Texas Neurology Consultants, Round Rock, Texas
- Italy (5):
  - Casa di Cura villa Margherita (Neurologia), Arcugnano
  - Centro Ricerche San Raffaele, Cassino
  - Agine Research Center, University Foundahon Chica-Pescara, Behavioral Neurology and Movement Disorders Unit, Chieti
  - Neurologia, Policlinico Tor Vergata, Rome
  - IRCCS San Raffaele Pisana,Clinical Trial Center, Rome

REFERENCES:
- [Derived] Stocchi F, Peckham EL, De Pandis MF, Sciarappa K, Kleiman R, Agbo F, Olanow CW, Blum D, Navia B. A Randomized Thorough QT Study of Apomorphine Sublingual Film in Patients With Parkinson's Disease. Clin Pharmacol Drug Dev. 2022 Sep;11(9):1068-1077. doi: 10.1002/cpdd.1147. Epub 2022 Jul 28. PMID 35899977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Parkinson's disease (PD) complicated by motor fluctuations ('OFF' episodes) were recruited in 13 study sites in Italy and the United States, starting April 2017. The study was completed in December 2017. Approval was obtained from the Enrollment Adjudication Committee and Sponsor prior to enrollment of each patient.
Pre-assignment Details: Dose Titration Phase: individual responses to single doses of APL 130277 were evaluated at 5 mg increments up to 40 mg and then 10 mg increments up to 60 mg until a full 'ON' was achieved. If tolerated, patients were titrated to a supratherapeutic dose (up to 60 mg) which was 1 or 2 levels above the initial dose producing an 'ON' response.
Groups:
- APL-130277, Then Placebo, Then Moxifloxacin: Sequence 1: Participants first received APL-130277. After a 3-day washout period, they then received Placebo. After a 3-day washout period, they then received Moxifloxacin.
- Placebo, Then Moxifloxacin, Then APL-130277: Sequence 2: Participants first received Placebo. After a 3-day washout period, they then received Moxifloxacin. After a 3-day washout period, they then received APL-130277.
- Moxifloxacin, Then APL-130277, Then Placebo: Sequence 3: Participants first received Moxifloxacin. After a 3-day washout period, they then received APL-130277. After a 3-day washout period, they then received Placebo.
- Moxifloxacin, Then Placebo, Then APL-130277: Sequence 4: Participants first received Moxifloxacin. After a 3-day washout period, they then received Placebo. After a 3-day washout period, they then received APL-130277.
- APL-130277, Then Moxifloxacin, Then Placebo: Sequence 5: Participants first received APL-130277. After a 3-day washout period, they then received Moxifloxacin. After a 3-day washout period, they then received Placebo.
- Placebo, Then APL-130277, Then Moxifloxacin: Sequence 6: Participants first received Placebo. After a 3-day washout period, they then received APL-130277. After a 3-day washout period, they then received Moxifloxacin.
- Sequence Not Assigned: Sequence Not Assigned: Participants not randomized to a treatment sequence.
Period: Titration Period
Arm/Group | APL-130277, Then Placebo, Then Moxifloxacin | Placebo, Then Moxifloxacin, Then APL-130277 | Moxifloxacin, Then APL-130277, Then Placebo | Moxifloxacin, Then Placebo, Then APL-130277 | APL-130277, Then Moxifloxacin, Then Placebo | Placebo, Then APL-130277, Then Moxifloxacin | Sequence Not Assigned
Started | 7 | 7 | 7 | 6 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 6 | 7 | 7 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Exclusion Criteria Met | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Pre-Intervention
Arm/Group | APL-130277, Then Placebo, Then Moxifloxacin | Placebo, Then Moxifloxacin, Then APL-130277 | Moxifloxacin, Then APL-130277, Then Placebo | Moxifloxacin, Then Placebo, Then APL-130277 | APL-130277, Then Moxifloxacin, Then Placebo | Placebo, Then APL-130277, Then Moxifloxacin | Sequence Not Assigned
Started | 7 | 7 | 7 | 6 | 7 | 7 | 0
Completed | 6 | 7 | 7 | 6 | 7 | 7 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: First Intervention
Arm/Group | APL-130277, Then Placebo, Then Moxifloxacin | Placebo, Then Moxifloxacin, Then APL-130277 | Moxifloxacin, Then APL-130277, Then Placebo | Moxifloxacin, Then Placebo, Then APL-130277 | APL-130277, Then Moxifloxacin, Then Placebo | Placebo, Then APL-130277, Then Moxifloxacin | Sequence Not Assigned
Started | 6 | 7 | 7 | 6 | 7 | 7 | 0
Completed | 6 | 7 | 7 | 6 | 7 | 7 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: First Washout
Arm/Group | APL-130277, Then Placebo, Then Moxifloxacin | Placebo, Then Moxifloxacin, Then APL-130277 | Moxifloxacin, Then APL-130277, Then Placebo | Moxifloxacin, Then Placebo, Then APL-130277 | APL-130277, Then Moxifloxacin, Then Placebo | Placebo, Then APL-130277, Then Moxifloxacin | Sequence Not Assigned
Started | 6 | 7 | 7 | 6 | 7 | 7 | 0
Completed | 6 | 7 | 7 | 6 | 7 | 7 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | APL-130277, Then Placebo, Then Moxifloxacin | Placebo, Then Moxifloxacin, Then APL-130277 | Moxifloxacin, Then APL-130277, Then Placebo | Moxifloxacin, Then Placebo, Then APL-130277 | APL-130277, Then Moxifloxacin, Then Placebo | Placebo, Then APL-130277, Then Moxifloxacin | Sequence Not Assigned
Started | 6 | 7 | 7 | 6 | 7 | 7 | 0
Completed | 6 | 7 | 7 | 6 | 7 | 7 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Washout
Arm/Group | APL-130277, Then Placebo, Then Moxifloxacin | Placebo, Then Moxifloxacin, Then APL-130277 | Moxifloxacin, Then APL-130277, Then Placebo | Moxifloxacin, Then Placebo, Then APL-130277 | APL-130277, Then Moxifloxacin, Then Placebo | Placebo, Then APL-130277, Then Moxifloxacin | Sequence Not Assigned
Started | 6 | 7 | 7 | 6 | 7 | 7 | 0
Completed | 6 | 7 | 7 | 6 | 7 | 7 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | APL-130277, Then Placebo, Then Moxifloxacin | Placebo, Then Moxifloxacin, Then APL-130277 | Moxifloxacin, Then APL-130277, Then Placebo | Moxifloxacin, Then Placebo, Then APL-130277 | APL-130277, Then Moxifloxacin, Then Placebo | Placebo, Then APL-130277, Then Moxifloxacin | Sequence Not Assigned
Started | 6 | 7 | 7 | 6 | 7 | 7 | 0
Completed | 6 | 7 | 7 | 6 | 7 | 7 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: APL-130277 (Titration): Patients who completed the Dose Titration Phase in Period 1 (N=41) were eligible to proceed to randomization in the crossover phase (Period 2). One patient discontinued prior to receiving any study medication; therefore, a total of 40 patients were dosed with study medication in the crossover phase (Period 2)
Groups:
- Overall (Cross-Over): Patients who successfully completed the Dose Titration Phase of the study were randomized to 1 of 6 treatment sequences in the single-dose Randomized Crossover Assessment Phase. Following confirmation by both the Investigator and the patient that the patient was in the 'OFF' state, the patient was dosed according to the patient's random treatment assignment with
  1. APL-130277 at the dose determined in the Dose Titration Phase; OR
  2. Matched placebo APL-130277; OR
  3. A single 400 mg dose of moxifloxacin. Patients were randomized in equal numbers to 6 possible sequences of the above 3 study treatments determined by a 3-way balanced crossover design.
  There was a 3-day washout period between treatment period dosing visits. Dosing of APL-130277 and placebo was double-blinded, and dosing of moxifloxacin was open-label.
Arm/Group | Overall (Cross-Over)
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
  Italy | 16
Time Since Diagnosis of PD [Mean (Standard Deviation); unit: years] | 8.30 (4.322)
Presence of a Rest Tremor at the Time of Diagnosis [Number; unit: participants]
  yes | 27
  no | 13
Time Since Initiationof L-dopa Treatment [Mean (Standard Deviation); unit: years] | 6.20 (4.502)
Time Since Motor Fluctuations Started [Mean (Standard Deviation); unit: years] | 5.05 (3.811)
Type of "OFF" Episode Experienced [Number; unit: participants]
  Morning akinesia | 6
  Wearing-off | 31
  Sudden-off | 1
  Dose failure | 1
  Delayed "ON" | 0
  Other | 1
Number of "OFF" Episodes/Day [Number; unit: "OFF" Episodes/day]
  zero | 1
  one | 0
  two | 3
  three | 14
  four | 12
  five | 9
  six | 1
Typical Length of "OFF" Episode [Mean (Standard Deviation); unit: hours] | 1.30 (0.915)
Total Daily L-Dopa Dose [Mean (Standard Deviation); unit: mg] | 620.5 (273.05)

OUTCOME MEASURES:

1. Primary Outcome: Time-Matched Change From Baseline in QTc, Placebo-Adjusted and Corrected for Heart Rate Based on the Fridericia Correction Method (QTcF) Using Delta Delta Method (ΔΔQTcF): Comparison Between APL-130277 and Placebo (Central Tendency Analysis)
Description: For the primary central tendency analysis, the changes from baseline (ΔQTcF) were compared between APL-130277 and placebo (ΔΔQTcF). Baseline was defined as the mean of the 9 ECGs (3 sets of triplicate ECGs) recorded at baseline (P1V1). In case any of the 9 ECGs were missing, the baseline was defined as the mean of the available baseline values. The post-dose ECGs were evaluated at 15, 30, 45 and 60 minutes (mins) and 2, 3 and 4 hours post-dose at each of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase. For each of the time points, an average value was calculated based on the 3 (or all available) ECGs. These average values were used in all change from baseline calculations.
Time Frame: Baseline to 15, 30, 45, 60 mins and 2, 3, and 4 hours post-dose for each of the 3 treatment period dosing visits.
Population: The ECG Population included all randomized patients who had evaluable baseline 12-lead ECG (Holter) data at P1V1 and at least one evaluable post-dose 12-lead ECG (Holter) assessment during the Randomized Crossover Assessment Phase.
  Please Note: The pre-specified primary comparison was between APL-130277 and Placebo.
Measure: Least Squares Mean (Standard Error); unit: msec
Groups:
- APL-130277 (Cross-over): Patients who received a single dose of APL-130277 (as determined in the Dose Titration Phase) in 1 of the 3 treatment period dosing visits during the Randomized Assessment Crossover Phase.
- Placebo (Cross-over): Patients who received a single dose of placebo in 1 of the 3 treatment period dosing visits during the Randomized Assessment Crossover Phase.
Arm/Group | APL-130277 (Cross-over) | Placebo (Cross-over)
Number analyzed (Participants) | 40 | 40
msec
  15 mins post-dose | 0.2 (1.98) | -3.7 (1.97)
  30 mins post-dose | 0.3 (1.98) | -2.7 (1.97)
  45 mins post-dose | 0.0 (1.98) | -3.7 (1.97)
  60 mins post-dose | 2.7 (1.98) | -3.5 (1.97)
  2 hours post-dose | 1.8 (1.98) | -3.0 (1.97)
  3 hours post-dose | 0.1 (1.98) | -1.6 (1.98)
  4 hours post-dose | -0.9 (1.98) | -0.2 (1.98)
Statistical Analysis 1: Comparison: APL-130277 (Cross-over) vs Placebo (Cross-over); 15 mins post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcF approach. The mixed model for repeated measurements (MMRM) included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcF as a covariate. The patient nested within sequence was included as a random effect; Test type: Non-Inferiority — For each post-dose time point, change from baseline (ΔQTcF) was compared between APL-130277 and placebo (ΔΔQTcF). The hypothesis of no clinical difference was accepted, if all upper limits of the two-sided 90% confidence intervals (CIs) for APL-130277 versus placebo fell below 10 msec; Least Square (LS) Mean Difference = 4.0, 90% CI 2-sided [0.5 to 7.4], Standard Error of Mean 2.11
Statistical Analysis 2: Comparison: APL-130277 (Cross-over) vs Placebo (Cross-over); 30 mins post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcF approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcF as a covariate. The patient nested within sequence was included as a random effect; Test type: Non-Inferiority — For each post-dose time point, change from baseline (ΔQTcF) was compared between APL-130277 and placebo (ΔΔQTcF). The hypothesis of no clinical difference was accepted, if all upper limits of the two-sided 90% CIs for APL-130277 versus placebo fell below 10 msec; Least Square (LS) Mean difference = 3.0, 90% CI 2-sided [-0.5 to 6.5], Standard Error of Mean 2.11
Statistical Analysis 3: Comparison: APL-130277 (Cross-over) vs Placebo (Cross-over); 45 mins post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcF approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcF as a covariate. The patient nested within sequence was included as a random effect; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least Square (LS) Mean Difference = 3.7, 90% CI 2-sided [0.2 to 7.2], Standard Error of Mean 2.11
Statistical Analysis 4: Comparison: APL-130277 (Cross-over) vs Placebo (Cross-over); 60 mins post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcF approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcF as a covariate. The patient nested within sequence was included as a random effect; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least Square (LS) Mean Difference = 6.2, 90% CI 2-sided [2.7 to 9.7], Standard Error of Mean 2.11
Statistical Analysis 5: Comparison: APL-130277 (Cross-over) vs Placebo (Cross-over); 2 hours post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcF approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcF as a covariate. The patient nested within sequence was included as a random effect; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least Square (LS) Mean Difference = 4.8, 90% CI 2-sided [1.3 to 8.3], Standard Error of Mean 2.11
Statistical Analysis 6: Comparison: APL-130277 (Cross-over) vs Placebo (Cross-over); 3 hours post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcF approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcF as a covariate. The patient nested within sequence was included as a random effect; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least Square (LS) Mean Difference = 1.8, 90% CI 2-sided [-1.7 to 5.3], Standard Error of Mean 2.12
Statistical Analysis 7: Comparison: APL-130277 (Cross-over) vs Placebo (Cross-over); 4 hours post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcF approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcF as a covariate. The patient nested within sequence was included as a random effect; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least Sqaure (LS) Mean Difference = -0.7, 90% CI [-4.2 to 2.8], Standard Error of Mean 2.12

2. Secondary Outcome: Cmax of Apomorphine and Apomorphine Sulfate (Metabolite) Following the Administration of APL-130277
Description: The maximum observed plasma concentration (Cmax) for apomorphine and apomorphine sulfate (metabolite) was determined in patients treated with APL-130277. Pharmacokinetic (PK) parameters were derived using a non-compartmental analysis method. Bioanalysis of apomorphine and apomorphine-sulfate plasma concentration were measured using a validated liquid chromatography-tandem mass spectrometry (LC/MS-MS) method. The calibration range was 0.0200 nanograms per milliliter (ng/mL) to 20.0 ng/mL apomorphine and 10.0 to 1000 ng/mL apomorphine sulfate (metabolite). PK assessments were performed at each period of the Randomized Crossover Assessment Phase (at P1V1, P2V2 and P3V3) and results are presented for each of the APL-130277 doses administered (as determined for each patient during the Dose Titration Phase).
Time Frame: Blood samples for PK assessments were taken prior to dosing and at 0.5, 0.75, 1, 2, and 4 hours post-dose.
Population: The PK population included all patients with at least one PK evaluation. Only patients with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 10 mg APL-130277 PK Subset: Patients who received a single dose of 10 mg APL-130277 (as determined in the Dose Titration Phase) in 1 of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
- 15mg AP:-130277 PK Subset: Patients who received a single dose of 15 mg APL-130277 (as determined in the Dose Titration Phase) in 1 of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
- 20 mg AP:-130277 PK Subset: Patients who received a single dose of 20 mg APL-130277 (as determined in the Dose Titration Phase) in 1 of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
- 25 mg APL-130277 PK Subset: Patients who received a single dose of 25 mg APL-130277 (as determined in the Dose Titration Phase) in 1 of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
- 35 mg APL-130277 PK Subset: Patients who received a single dose of 35 mg APL-130277 (as determined in the Dose Titration Phase) in 1 of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
- 50 mg AP:-130277 PK Subset: Patients who received a single dose of 50 mg APL-130277 (as determined in the Dose Titration Phase) in 1 of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
Arm/Group | 10 mg APL-130277 PK Subset | 15mg AP:-130277 PK Subset | 20 mg AP:-130277 PK Subset | 25 mg APL-130277 PK Subset | 35 mg APL-130277 PK Subset | 50 mg AP:-130277 PK Subset
Number analyzed (Participants) | 14 | 4 | 15 | 2 | 3 | 1
ng/mL
  Apomorphine | 5.14 (3.28) | 6.57 (1.22) | 4.23 (2.81) | 4.16 (2.54) | 9.29 (9.97) | 4.61 (NA) — only 1 subject analyzed- cmax was determined for one patient so calculation of standard deviation was not applicable
  Apomorphine sulfate | 220 (77.4) | 319 (97.9) | 377 (82.0) | 446 (46.7) | 458 (12.7) | 1420 (NA) — only 1 subject analyzed- cmax was determined for one patient so calculation of standard deviation was not applicable

3. Secondary Outcome: Tmax of Apomorphine and Apomorphine Sulfate (Metabolite) Following the Administration of APL-130277
Description: The time of maximum observed plasma concentration (Tmax) for apomorphine and apomorphine sulfate (metabolite) was determined in patients treated with APL-130277. PK parameters were derived using a non-compartmental analysis method. Bioanalysis of apomorphine and apomorphine-sulfate plasma concentration were measured using a validated LC/MS-MS method. The calibration range was 0.0200 ng/mL to 20.0 ng/mL apomorphine and 10.0 to 1000 ng/mL apomorphine sulfate. PK assessments were performed at each period of the Randomized Crossover Assessment Phase (at P1V1, P2V2 and P3V3) and results are presented for each of the APL-130277 doses administered (as determined for each patient during the Dose Titration Phase).
Time Frame: Blood samples for PK assessments were taken prior to dosing and at 0.5, 0.75, 1, 2, and 4 hours post-dose.
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Groups:
- 15 mg APL-130277 PK Subset: Patients who received a single dose of 15 mg APL-130277 (as determined in the Dose Titration Phase) in 1 of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
- 20 mg APL-130277 PK Subset: Patients who received a single dose of 20 mg APL-130277 (as determined in the Dose Titration Phase) in 1 of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
- 50 mg APL-130277 PK Subset: Patients who received a single dose of 50 mg APL-130277 (as determined in the Dose Titration Phase) in 1 of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
Arm/Group | 10 mg APL-130277 PK Subset | 15 mg APL-130277 PK Subset | 20 mg APL-130277 PK Subset | 25 mg APL-130277 PK Subset | 35 mg APL-130277 PK Subset | 50 mg APL-130277 PK Subset
Number analyzed (Participants) | 14 | 4 | 15 | 2 | 3 | 1
hours
  Apomorphine | 0.75 [0.50 to 1.02] | 0.75 [0.50 to 0.75] | 1.00 [0.50 to 2.07] | 1.50 [1.00 to 2.00] | 0.58 [0.50 to 0.88] | 0.78 [NA to NA] — Tmax was determined for one patient so calculation of standard deviation was not applicable
  Apomorphne sulfate | 2.00 [1.00 to 4.00] | 1.52 [0.75 to 2.17] | 2.00 [0.50 to 2.07] | 1.50 [1.00 to 2.00] | 2.13 [1.00 to 4.08] | 0.52 [NA to NA] — Tmax was determined for one patient so calculation of standard deviation was not applicable

4. Secondary Outcome: AUClast of Apomorphine and Apomorphine Sulfate (Metabolite) Following the Administration of APL-130277
Description: The area under the concentration-time curve from time of dosing to the last measurable point (AUClast) for apomorphine and apomorphine sulfate (metabolite) was determined in patients treated with APL-130277. PK parameters were derived using a non-compartmental analysis method. Bioanalysis of apomorphine and apomorphine-sulfate plasma concentration were measured using a validated LC/MS-MS method. The calibration range was 0.0200 ng/mL to 20.0 ng/mL apomorphine and 10.0 to 1000 ng/mL apomorphine sulfate. PK assessments were performed at each period of the Randomized Crossover Assessment Phase (at P1V1, P2V2 and P3V3) and results are presented for each of the APL-130277 doses administered (as determined for each patient during the Dose Titration Phase).
Time Frame: Blood samples for PK assessments were taken prior to dosing and at 0.5, 0.75, 1, 2, and 4 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 10 mg APL-130277 PK Subset | 15 mg APL-130277 PK Subset | 20 mg APL-130277 PK Subset | 25 mg APL-130277 PK Subset | 35 mg APL-130277 PK Subset | 50 mg APL-130277 PK Subset
Number analyzed (Participants) | 14 | 4 | 15 | 2 | 3 | 1
h*ng/mL
  Apomorphine | 7.70 (4.15) | 9.39 (3.31) | 7.55 (3.81) | 7.84 (0.975) | 12.1 (6.63) | 10.9 (NA) — AUClast was determined for one patient so calculation of standard deviation was not applicable.
  Apomorphine sulfate | 558 (161) | 734 (155) | 861 (147) | 870 (108) | 979 (127) | 1980 (NA) — AUClast was determined for one patient so calculation of standard deviation was not applicable.

5. Secondary Outcome: Number of Patients With Treatment-Emergent Adverse Events (TEAEs)
Description: AE definition: any untoward medical occurrence in a clinical trial participant. Serious AE definition: an AE that is fatal, life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in permanent (persistent) disability/incapacity, is a congenital anomaly/birth defect or is an important medical event. Severity of AEs were classified as: mild: causes no limitation of usual activities, moderate: causes some limitation of usual activities; or severe: prevents or severely limits usual activities. The investigator assessed AEs for relatedness to study medication. TEAEs were defined as all AEs that started on or after the first dose of study medication (APL-130277, moxifloxacin or placebo). Results are presented for TEAEs during the Randomized Crossover Assessment Phase.
Time Frame: From first dose of study medication up to last study visit for Randomized Crossover Assessment Phase, approximately up to 2 weeks
Population: The Crossover Phase Safety Population consisted of all patients who were randomized and received at least one post-randomization dose of study medication (APL-130277, moxifloxacin or placebo) during the Randomized Crossover Assessment Phase.
Measure: Number; unit: participants
Groups:
- Placebo (Crossover): Patients who received a single dose of placebo in 1 of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
- Moxifloxacin (Crossover): Patients who received a single dose of 400 mg moxifloxacin in 1 of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
Arm/Group | APL-130277 (Cross-over) | Placebo (Crossover) | Moxifloxacin (Crossover)
Number analyzed (Participants) | 40 | 40 | 40
participants
  Any TEAE | 13 | 6 | 4
  Drug-related TEAE | 12 | 2 | 0
  Severe TEAE | 1 | 0 | 0
  Serious TEAE | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0

6. Secondary Outcome: ECG Assessments: Mean Change From Baseline to Post-Baseline Value for QTcB Interval During Randomized Crossover Assessment Phase
Description: QTcB was defined as QT interval corrected with Bazett's method. QT was defined as time between start of Q wave and end of T wave. QTcB was determined during continuous 12-lead ECG (Holter) monitoring at each of the 3 treatment period dosing visits at pre-specified timepoints post-dose. Baseline was defined as the mean of the 9 ECGs (3 sets of triplicate ECGs) recorded at baseline (pre-dose P1V1). In case any of the 9 ECGs were missing, the baseline was defined as the mean of the available baseline values. The post-dose ECGs were evaluated at 15, 30, 45 and 60 mins and 2, 3 and 4 hours post-dose at each of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase. For each of the time points, an average value was calculated based on the 3 (or all available) ECGs. Results are presented for the mean change from baseline at each pre-specified post-dose timepoint.
Time Frame: Baseline and at 15, 30, 45, 60 minutes and 2, 3, and 4 hours post-dose for each of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
Population: The ECG Population included all randomized patients who had evaluable baseline 12-lead ECG (Holter) data at P1V1 and at least one evaluable post-dose 12-lead ECG (Holter) assessment during the Randomized Crossover Assessment Phase.
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | APL-130277 (Cross-over) | Placebo (Crossover) | Moxifloxacin (Crossover)
Number analyzed (Participants) | 40 | 40 | 40
msec
  15 mins post-dose | 2.7 (2.24) | -1.7 (2.22) | -2.5 (2.23)
  30 mins post-dose | 1.9 (2.24) | -0.7 (2.22) | 1.4 (2.23)
  45 mins post-dose | 0.1 (2.24) | -3.2 (2.22) | 7.8 (2.23)
  60 mins post-dose | -0.1 (2.24) | -3.3 (2.22) | 8.4 (2.23)
  2 hours post-dose | 4.7 (2.24) | -0.4 (2.22) | 11.1 (2.25)
  3 hours post-dose | 7.2 (2.24) | 2.7 (2.24) | 12.8 (2.23)
  4 hours post-dose | 8.1 (2.24) | 5.5 (2.24) | 12.1 (2.23)
Statistical Analysis 1: Comparison: APL-130277 (Cross-over) vs Placebo (Crossover); Test type: Non-Inferiority — 15 mins post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcB approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcB as a covariate. The patient nested within sequence was included as a random effect; Least Square (LS) Mean Difference = 4.4, 90% CI 2-sided [0.3 to 8.6], Standard Error of Mean 2.54
Statistical Analysis 2: Comparison: APL-130277 (Cross-over) vs Placebo (Crossover); Test type: Non-Inferiority — 30 mins post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcB approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcB as a covariate. The patient nested within sequence was included as a random effect; Least Square (LS) Mean Difference = 2.5, 90% CI 2-sided [-1.6 to 6.7], Standard Error of Mean 2.54
Statistical Analysis 3: Comparison: APL-130277 (Cross-over) vs Placebo (Crossover); Test type: Non-Inferiority — 45 mins post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcB approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcB as a covariate. The patient nested within sequence was included as a random effect; Least Square (LS) Mean Difference = 3.2, 90% CI 2-sided [-0.9 to 7.4], Standard Error of Mean 2.54
Statistical Analysis 4: Comparison: APL-130277 (Cross-over) vs Placebo (Crossover); Test type: Non-Inferiority — 60 mins post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcB approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcB as a covariate. The patient nested within sequence was included as a random effect; Least Square (LS) Mean Difference = 3.3, 90% CI 2-sided [-0.9 to 7.5], Standard Error of Mean 2.54
Statistical Analysis 5: Comparison: APL-130277 (Cross-over) vs Placebo (Crossover); Test type: Non-Inferiority — 2 hours post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcB approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcB as a covariate. The patient nested within sequence was included as a random effect; Least Square (LS) Mean Difference = 5.0, 90% CI 2-sided [0.8 to 9.2], Standard Error of Mean 2.54
Statistical Analysis 6: Comparison: APL-130277 (Cross-over) vs Placebo (Crossover); Test type: Non-Inferiority — 3 hours post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcB approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcB as a covariate. The patient nested within sequence was included as a random effect; Least Square (LS) Mean Difference = 4.6, 90% CI 2-sided [0.4 to 8.8], Standard Error of Mean 2.55
Statistical Analysis 7: Comparison: APL-130277 (Cross-over) vs Placebo (Crossover); Test type: Non-Inferiority — 4 hours post-dose: time-matched, baseline-corrected comparison between APL-130277 and placebo using the ΔΔQTcB approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcB as a covariate. The patient nested within sequence was included as a random effect; Least Square (LS) Mean Differeence = 2.6, 90% CI 2-sided [-1.6 to 6.9], Standard Error of Mean 2.56

7. Secondary Outcome: Mean Change From Pre-Dose to Post-Baseline Value in the Movement Disorders Society Unified Parkinson's Disease Rating Scale Part III Motor Examination (MDS-UPDRS Part III) Score During the Dose Titration Phase
Description: The Motor Function section (Part III) of the MDS-UPDRS was administered by the Investigator, and included 33 scores based on 18-items, each anchored with 5 responses: 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range was from 0 to 132, with a lower score indicating better motor function and a higher score indicating more severe motor symptoms.
  The least squares mean change in the MDS-UPDRS Part III score from pre-dose to 30, 60 and 90 minutes post-dose during the Dose Titration Phase at the highest tolerated APL-130277 dose level (indicated as Day 2) and the lowest APL-130277 dose resulting in a full 'ON' (indicated as Day 1) are presented.
Time Frame: Baseline (pre-dose) and at 30, 60 and 90 minutes after dosing during the Dose Titration Phase.
Population: The Efficacy Population included all patients who had efficacy assessments at the lowest dose level resulting in a full 'ON' and at a higher dose level during the Dose Titration Phase.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- APL-130277 (Titration): Patients were titrated to an effective and tolerable dose of APL-130277. Patients were dosed with increasing doses of APL 130277 starting with 10 mg at TV 1 up to a maximum of 60 mg. Patients who did not achieve a complete and full 'ON' response with the 10 mg APL 130277 dose at TV1 restarted their normal PD medications and were asked to return to the clinic the next business day for TV2, to assess the next highest dose. The evaluation continued sequentially with 15 mg (TV2), 20 mg (TV3), 25 mg (TV4), 30 mg (TV5), 35 mg (TV6), 40 mg (TV7), 50 mg (TV8), and 60 mg (TV9) doses of APL-130277 until a full 'ON' state was achieved. If tolerated, patients were titrated to a supratherapeutic dose (up to 60 mg) which was 1 or 2 levels above the initial dose producing an 'ON' response. If the patient was unable to tolerate 1 or either of the 2 additional dose levels after reaching a full "ON" state patients were randomized to the previous tolerable dose.
Arm/Group | APL-130277 (Titration)
Number analyzed (Participants) | 35
units on a scale
  30 mins post-dose (day 1) | -21.1 (1.79)
  30 mins post-dose (day 2) | -26.7 (1.78)
  60 mins post-dose (day 1) | -26.3 (1.46)
  60 mins post-dose (day 2) | -31.3 (1.72)
  90 mins post-dose (day 1) | -25.2 (1.43)
  90 mins post-dose (day 2) | -28.9 (1.68)

8. Secondary Outcome: Median Time to 'ON' During the Dose Titration Phase
Description: The time to 'ON' was calculated as minutes from the time when the patient received APL-130277 until the time the patient turned fully 'ON', as assessed by the Investigator. Data was censored at 90 minutes.
  The median time to a full 'ON' response during the Dose Titration Phase following the highest tolerated APL-130277 dose level (indicated as Day 2) and the lowest APL-130277 dose resulting in a full 'ON' (indicated as Day 1) are presented. The median time to 'ON' on Day 1 and Day 2 was calculated using the Kaplan-Meier method.
Time Frame: Time of dosing up to 90 minutes post-dose during the Dose Titration Phase.
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | APL-130277 (Titration)
Number analyzed (Participants) | 35
minutes
  Day 1 | 30 [22 to 45]
  Day 2 | 30 [22 to 60]

9. Secondary Outcome: Median Duration of 'ON' During the Dose Titration Phase
Description: The duration of 'ON' was calculated as minutes from the time when the patient turned fully 'ON' until the time when the patient turned 'OFF', as assessed by the Investigator. If the patient did not turn fully 'ON' within 90 minutes the duration of 'ON' was defined as zero minutes. If the patient turned fully 'ON' and did not turn 'OFF' by 90 minutes, the data was censored at 90 minutes minus the time when the patient turned fully 'ON'.
  The median duration of a full 'ON' response during the Dose Titration Phase following the highest tolerated APL-130277 dose level (indicated as Day 2) and the lowest APL-130277 dose resulting in a full 'ON' (indicated as Day 1) are presented. The median duration of 'ON' on Day 1 and Day 2 was calculated using the Kaplan-Meier method.
Time Frame: Time of dosing up to 90 minutes post-dose during the Dose Titration Phase.
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: minutess
Arm/Group | APL-130277 (Titration)
Number analyzed (Participants) | 35
minutess
  Day 1 | NA [NA to NA] — The median duration and inter-quartile range could not be estimated because approximately 90% of patients were censored (i.e. still 'ON' at last observation) on both days
  Day 2 | NA [NA to NA] — The median duration and inter-quartile range could not be estimated because approximately 90% of patients were censored (i.e. still 'ON' at last observation) on both days

10. Primary Outcome: Time-Matched Change From Baseline in QTc, Placebo-Adjusted and Corrected for Heart Rate Based on QTcF Using ΔΔQTcF: Comparison Between Moxifloxacin and Placebo (Assay Sensitivity Analysis)
Description: For the assay sensitivity analysis in support of the primary central tendency analysis, the changes from baseline (ΔQTcF) were compared between moxifloxacin (positive control) and placebo (ΔΔQTcF). Baseline was defined as the mean of the 9 ECGs (3 sets of triplicate ECGs) recorded at baseline (P1V1). In case any of the 9 ECGs were missing, the baseline was defined as the mean of the available baseline values. The post-dose ECGs were evaluated at 60 mins and 2, 3 and 4 hours post-dose for each of the 3 treatment period dosing visits in the Randomized Crossover Assessment Phase. For each of the time points, an average value was calculated based on the 3 (or all available) ECGs. These average values were used in all change from baseline calculations.
Time Frame: Baseline to 60 mins and 2, 3, and 4 hours post-dose for each of the 3 treatment period dosing visits.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Moxifloxacin (Crossover) | Placebo (Cross-over)
Number analyzed (Participants) | 40 | 40
msec
  60 mins post-dose | 6.5 (1.98) | -3.5 (1.97)
  2 hours post-dose | 9.3 (1.99) | -3.0 (1.97)
  3 hours post-dose | 9.3 (1.98) | -1.6 (1.98)
  4 hours post-dose | 8.8 (1.98) | -0.2 (1.98)
Statistical Analysis 1: Comparison: Moxifloxacin (Crossover) vs Placebo (Cross-over); 60 mins post-dose: time-matched, baseline-corrected comparison between moxifloxacin and placebo using the ΔΔQTcF approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcF as a covariate. The patient nested within sequence was included as a random effect; Test type: Non-Inferiority — The hypothesis of assay sensitivity(difference in QTcF time between moxifloxacin and placebo)was evaluated by observing if any of the 4 post-dose evaluation time points had a one-sided(Bonferroni-corrected)95% lower confidence limit which was equal to, or exceeded, 5 msec; Least Square (LS) Mean Difference = 10.0, 90% CI 2-sided [5.3 to 14.8], Standard Error of Mean 2.11
Statistical Analysis 2: Comparison: Moxifloxacin (Crossover) vs Placebo (Cross-over); 2 hours post-dose: time-matched, baseline-corrected comparison between moxifloxacin and placebo using the ΔΔQTcF approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcF as a covariate. The patient nested within sequence was included as a random effect; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; Least Square (LS) Mean Difference = 12.3, 90% CI 2-sided [7.5 to 17.1], Standard Error of Mean 2.12
Statistical Analysis 3: Comparison: Moxifloxacin (Crossover) vs Placebo (Cross-over); 3 hours post-dose: time-matched, baseline-corrected comparison between moxifloxacin and placebo using the ΔΔQTcF approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcF as a covariate. The patient nested within sequence was included as a random effect; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; Least Square (LS) Mean Difference = 10.9, 90% CI 2-sided [6.1 to 15.7], Standard Error of Mean 2.12
Statistical Analysis 4: Comparison: Moxifloxacin (Crossover) vs Placebo (Cross-over); 4 hours post-dose: time-matched, baseline-corrected comparison between moxifloxacin and placebo using the ΔΔQTcF approach. The MMRM included region, gender, planned sequence, period, treatment, time, and interaction between treatment and time as fixed factors, and baseline QTcF as a covariate. The patient nested within sequence was included as a random effect; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; Least Square (LS) Mean Difference = 9.0, 90% CI 2-sided [4.2 to 13.8], Standard Error of Mean 2.12

11. Secondary Outcome: ECG Assessments: Mean Change From Baseline to Post-Baseline Value for Heart Rate During Randomized Crossover Assessment Phase
Description: Heart rate was determined during continuous 12-lead ECG (Holter) monitoring at each of the 3 treatment period dosing visits at pre-specified timepoints post-dose. Baseline was defined as the mean of the 9 ECGs (3 sets of triplicate ECGs) recorded at baseline (pre-dose P1V1). In case any of the 9 ECGs were missing, the baseline was defined as the mean of the available baseline values. The post-dose ECGs were evaluated at 15, 30, 45 and 60 mins and 2, 3 and 4 hours post-dose at each of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase. For each of the time points, an average value was calculated based on the 3 (or all available) ECGs. Results are presented for the mean change from baseline at each pre-specified post-dose timepoint.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | APL-130277 (Cross-over) | Placebo (Cross-over) | Moxifloxacin (Crossover)
Number analyzed (Participants) | 40 | 40 | 40
Beats per minute
  15 mins post-dose | 2.5 (1.31) | 2.1 (1.30) | 0.1 (1.31)
  30 mins post-dose | 1.5 (1.31) | 2.1 (1.30) | 0.5 (1.31)
  45 mins post-dose | 0.1 (1.31) | 0.8 (1.30) | 3.6 (1.31)
  60 mins post-dose | -3.0 (1.31) | 0.1 (1.30) | 1.8 (1.31)
  2 hours post-dose | 3.3 (1.31) | 2.8 (1.30) | 1.5 (1.32)
  3 hours post-dose | 7.6 (1.31) | 4.6 (1.31) | 3.3 (1.31)
  4 hours post-dose | 9.5 (1.31) | 6.2 (1.31) | 2.9 (1.31)

12. Secondary Outcome: ECG Assessments: Mean Change From Baseline to Post-Baseline Value for PR Interval During Randomized Crossover Assessment Phase
Description: PR interval was defined as time from the onset of the P wave to the start of the QRS complex. PR interval was determined during continuous 12-lead ECG (Holter) monitoring at each of the 3 treatment period dosing visits at pre-specified timepoints post-dose. Baseline was defined as the mean of the 9 ECGs (3 sets of triplicate ECGs) recorded at baseline (pre-dose P1V1). In case any of the 9 ECGs were missing, the baseline was defined as the mean of the available baseline values. The post-dose ECGs were evaluated at 15, 30, 45 and 60 mins and 2, 3 and 4 hours post-dose at each of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase. For each of the time points, an average value was calculated based on the 3 (or all available) ECGs. Results are presented for the mean change from baseline at each pre-specified post-dose timepoint.
Time Frame: Baseline (pre-dose P1V1) and at 15, 30, 45, 60 minutes and 2, 3, and 4 hours post-dose for each of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | APL-130277 (Cross-over) | Placebo (Cross-over) | Moxifloxacin (Crossover)
Number analyzed (Participants) | 40 | 40 | 40
msec
  15 mins post-dose | 0.4 (1.72) | -1.9 (1.71) | -1.1 (1.72)
  30 mins post-dose | -1.6 (1.73) | -0.2 (1.71) | -0.2 (1.72)
  45 mins post-dose | 1.2 (1.72) | 0.1 (1.71) | -1.1 (1.72)
  60 mins post-dose | 2.5 (1.72) | -0.3 (1.71) | 1.5 (1.72)
  2 hours post-dose | -0.2 (1.72) | -1.7 (1.71) | -0.1 (1.73)
  3 hours post-dose | -1.5 (1.73) | -2.2 (1.72) | 1.6 (1.72)
  4 hours post-dose | -3.7 (1.73) | -3.1 (1.72) | 0.8 (1.72)

13. Secondary Outcome: ECG Assessments: Mean Change From Baseline to Post-Baseline Value for QRS Interval During Randomized Crossover Assessment Phase
Description: QRS interval was defined as the time of QRS complex (Q, R, and S waves). QRS interval was determined during continuous 12-lead ECG (Holter) monitoring at each of the 3 treatment period dosing visits at pre-specified timepoints post-dose. Baseline was defined as the mean of the 9 ECGs (3 sets of triplicate ECGs) recorded at baseline (pre-dose P1V1). In case any of the 9 ECGs were missing, the baseline was defined as the mean of the available baseline values. The post-dose ECGs were evaluated at 15, 30, 45 and 60 mins and 2, 3 and 4 hours post-dose at each of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase. For each of the time points, an average value was calculated based on the 3 (or all available) ECGs. Results are presented for the mean change from baseline at each pre-specified post-dose timepoint.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | APL-130277 (Cross-over) | Placebo (Cross-over) | Moxifloxacin (Crossover)
Number analyzed (Participants) | 40 | 40 | 40
msec
  15 mins post-dose | -0.7 (0.94) | -1.2 (0.93) | -0.7 (0.94)
  30 mins post-dose | -0.4 (0.94) | -0.9 (0.93) | -0.1 (0.94)
  45 mins post-dose | -1.2 (0.94) | -0.1 (0.93) | -0.9 (0.94)
  60 mins post-dose | -0.8 (0.94) | -1.4 (0.93) | -0.4 (0.94)
  2 hours post-dose | 1.1 (0.94) | -1.3 (0.93) | -1.1 (0.95)
  3 hours post-dose | -0.2 (0.94) | -0.9 (0.94) | -1.0 (0.94)
  4 hours post-dose | 0.5 (0.94) | -0.6 (0.94) | 0.4 (0.94)

14. Secondary Outcome: ECG Assessments: Mean Change From Baseline to Post-Baseline Value for Uncorrected QT Interval During Randomized Crossover Assessment Phase
Description: Uncorrected QT interval was defined as time between start of Q wave and end of T wave. QT interval was determined during continuous 12-lead ECG (Holter) monitoring at each of the 3 treatment period dosing visits at pre-specified timepoints post-dose. Baseline was defined as the mean of the 9 ECGs (3 sets of triplicate ECGs) recorded at baseline (pre-dose P1V1). In case any of the 9 ECGs were missing, the baseline was defined as the mean of the available baseline values. The post-dose ECGs were evaluated at 15, 30, 45 and 60 mins and 2, 3 and 4 hours post-dose at each of the 3 treatment period dosing visits during the Randomized Crossover Assessment Phase. For each of the time points, an average value was calculated based on the 3 (or all available) ECGs. Results are presented for the mean change from baseline at each pre-specified post-dose timepoint.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | APL-130277 (Cross-over) | Placebo (Cross-over) | Moxifloxacin (Crossover)
Number analyzed (Participants) | 40 | 40 | 40
msec
  15 mins post-dose | -3.9 (3.05) | -7.1 (3.02) | -2.7 (3.04)
  30 mins post-dose | -2.2 (3.05) | -6.1 (3.02) | -0.7 (3.04)
  45 mins post-dose | 0.3 (3.05) | -4.2 (3.02) | -2.2 (3.04)
  60 mins post-dose | 8.3 (3.05) | -3.5 (3.02) | 3.5 (3.04)
  2 hours post-dose | -2.6 (3.05) | -7.6 (3.02) | 6.2 (3.07)
  3 hours post-dose | -12.0 (3.05) | -8.9 (3.04) | 3.0 (3.04)
  4 hours post-dose | -16.4 (3.05) | -10.1 (3.05) | 2.8 (3.04)

ADVERSE EVENTS:
Time Frame: Dose Titration Phase (up to 28 days): all AEs that started on/after the first dose of APL-130277 but before the first dose of study medication during the Randomized Crossover Assessment Phase. Randomized Crossover Assessment Phase (up to 18 days): all AEs that started on/after the first dose of study medication during the Crossover Phase up to end of study.
Description: All AEs were collected for each patient. Patients were queried in a non-leading manner, without specific prompting. TEAEs are presented for the Dose Titration Phase (APl-130277 [titration]) and for the Randomized Crossover Assessment Phase (APL-130277 [crossover], Placebo [crossover] and Moxifloxacin [crossover]).
Groups:
- APL-130277 (Cross-over): Patients who successfully completed the Dose Titration Phase of the study were randomized to 1 of 6 treatment sequences in the single-dose Randomized Crossover Assessment Phase. Following confirmation by both the Investigator and the patient that the patient was in the 'OFF' state, the patient was dosed according to the patient's random treatment assignment with
  1. APL-130277 at the dose determined in the Dose Titration Phase; OR
  2. Matched placebo APL-130277; OR
  3. A single 400 mg dose of moxifloxacin. Patients were randomized in equal numbers to 6 possible sequences of the above 3 study treatments determined by a 3-way balanced crossover design.
  There was a 3-day washout period between treatment period dosing visits. Dosing of APL-130277 and placebo was double-blinded, and dosing of moxifloxacin was open-label.
Arm/Group | APL-130277 (Titration) | APL-130277 (Cross-over) | Placebo (Crossover) | Moxifloxacin (Crossover)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 41/48 | 13/40 | 6/40 | 4/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APL-130277 (Titration) (N=48) | APL-130277 (Cross-over) (N=40) | Placebo (Crossover) (N=40) | Moxifloxacin (Crossover) (N=40)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 27 (35) | 4 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (9) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight descreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 12 (20) | 6 (6) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spontaneous penile erection (Reproductive system and breast disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Yawning (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hot Flush (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (5) | 1 (2) | 0 (0) | 2 (3)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT03187301/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT03187301/SAP_001.pdf